CLINICAL TRIAL: NCT04703842
Title: A Phase 1/2 Trial of the Safety and Efficacy of SRD-001 (AAV1/SERCA2a) in Subjects With Heart Failure With Reduced Ejection Fraction
Brief Title: Modulation of SERCA2a of Intra-myocytic Calcium Trafficking in Heart Failure With Reduced Ejection Fraction
Acronym: MUSIC-HFrEF1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sardocor Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRD-001-1001
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Congestive Heart Failure; Heart Failure, Systolic; Heart Failure; HFrEF - Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SRD-001 (Experimental): 3E13 or 4.5E13 vg; one-time intracoronary infusion
  Interventions: Biological: SRD-001
- Placebo (Placebo Comparator): One-time intracoronary infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: SRD-001 — AAV1/SERCA2a
  Arms: SRD-001
Drug: Placebo — SRD-001 matching placebo
  Arms: Placebo

SUMMARY:
It is believed that targeted SERCA2a enzyme replacement in HFrEF patients will correct defective intracellular Ca2+ hemostasis, resulting in improved cardiac contractile function and energetics which will, in turn, translate to improved clinical outcomes. Additionally, it is hypothesized that correcting SERCA2a dysfunction will also improve coronary blood flow through correction of the impaired endothelium-dependent nitric oxide-mediated vasodilatation observed in heart failure.

DETAILED DESCRIPTION:
MUSIC-HFrEF1 is an interventional study of SRD-001, an adeno-associated virus serotype 1 (AAV1) vector expressing the transgene for sarco(endo)plasmic reticulum Ca2+ ATPase 2a isoform (SERCA2a), in anti-AAV1 neutralizing antibody (NAb) negative subjects with ischemic or non-ischemic cardiomyopathy and New York Heart Association (NYHA) class III/IV symptoms of heart failure with reduced ejection fraction (HFrEF).

The Phase 1 trial is an open-label, uncontrolled study investigating two doses of SRD-001 at 3E13 and 4.5E13 viral genomes (vg) in 3-4 participants at each dose level.

The Phase 2 trial is a randomized, double-blind, placebo-controlled trial with prospective assignment to a single dose of either SRD-001 or placebo in a 1:1 ratio and a total sample size of N=50.

ELIGIBILITY:
Main Inclusion Criteria:

* Chronic ischemic or non-ischemic cardiomyopathy
* NYHA class III/IV
* LVEF ≤35%
* Guideline-directed medical therapy for heart failure; ICD

Main Exclusion Criteria:

* Restrictive cardiomyopathy, hypertrophic cardiomyopathy, acute myocarditis, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease or discrete left ventricular (LV) aneurysm
* Prior heart transplantation, left ventricular reduction surgery (LVRS), cardiomyoplasty, passive restraint device (e.g., CorCap™ Cardiac Support Device), mechanical circulatory support device (MCSD) or cardiac shunt
* Likely to receive cardiac resynchronization therapy, cardiomyoplasty, LVRS, conventional revascularization procedure or valvular repair in the 6 months following treatment
* Likely need for an immediate heart transplant or MCSD implant due to hemodynamic instability
* Inadequate hepatic and renal function
* Diagnosis of, or treatment for, any cancer within the last 5 years except for basal cell carcinoma or carcinomas in situ where surgical excision was considered curative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in symptomatic parameters | Baseline to Month 6 and Month 12
  New York Heart Association classification (I, II, III or IV)
Change from baseline in symptomatic parameters | Baseline to Month 6 and Month 12
  Quality of life as assessed by Kansas City Cardiomyopathy Questionnaire: 0-24, very poor to poor; 25-49, poor to fair; 50-74, fair to good; and 75-100, good to excellent
Change from baseline in physical parameter | Baseline to Month 6 and Month 12
  Distance walked during the 6MWT
Change from baseline in LV function/remodeling | Baseline to Month 6 and Month 12
  Left ventricular end systolic volume (LVESV) as assessed by echocardiography
Rate of recurrent events | Baseline to Month 6 and Month 12
  HF-related hospitalization, ambulatory worsening heart failure, all-cause death, MCSD and transplant
Rate of adverse events | 6 and 12 months
  Treatment-emergent adverse events

SECONDARY OUTCOMES:
Proportion of subjects who complete the trial | 12 months
  Those who complete the trial vs withdraw consent, are lost to follow-up, or withdrawn due to an AE or other reason
Concomitant medication use | 6 and 12 months
  Changes in heart failure related medications
Incidence of abnormal laboratory test results | Baseline to Month 6 and Month 12
  Hematologic, serum chemistries, NT-proBNP and troponin
Incidence of abnormal ECG results | Baseline to Month 6 and Month 12
  New arrhythmias
Incidence of abnormal physical examination findings | Baseline to Month 6 and Month 12
  Change from baseline in physical examination findings
Incidence of abnormal findings from interrogation of implantable cardioverter defibrillator | Baseline to Month 6 and Month 12
  New arrhythmias

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - San Diego Cardiac Center, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Washington University in Saint Louis, St Louis, Missouri
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No